CLINICAL TRIAL: NCT01441700
Title: A Comparative Study of Haemodynamic Changes Between Prone and Supine Emergence From Anaesthesia in Lumbar Disc Surgery
Brief Title: Prone Position Emergence From Anaesthesia in Lumbar Disc Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KVG Medical College and Hospital (Other)
Responsible Party: Principal Investigator, shivakumar m c, Assistant professor, KVG Medical College and Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMC/CT/1/2010; KVGMCH/CT/1/2010 (Other: KVGMCH)
Record Dates: First submitted 2011-09-24; First posted 2011-09-28 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2011-09

CONDITIONS: Haemodynamic Changes During During Emergence; Airway Response During Emergence; Monitor Disconnection During Emergence
Keywords: Prone emergence; supine emergence; coughing; haemodynamic stimulation; lumbar surgery
MeSH Terms: conditions — Cough | interventions — Prone Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prone position (Active Comparator)
  Interventions: Procedure: Prone and Supine emergence from anaesthesia
- Supine position (Active Comparator)
  Interventions: Procedure: Prone and Supine emergence from anaesthesia

INTERVENTIONS:
Procedure: Prone and Supine emergence from anaesthesia — Aims: The aim of this study was to compare haemodynamic changes and to evaluate the incidence of coughing, laryngospasm, loss of monitoring in patients undergoing lumbar disc surgery extubated in prone position and supine position. Settings and design: This open-level prospective randomized study was carried out in 50 patients who were admitted for elective lumbar surgery. Methods: The patients were randomly allocated to one of the two groups of 25 each at conclusion of surgery. First group was extubated in prone position and second in supine position at conclusion of surgery. Supine group patients were rolled back and prone group patients were left undisturbed. Extubation was done after complete reversal of neuromuscular block. Heart rates, Mean Arterial Pressure were noted at various points of time. Coughing, laryngospasm, vomiting, monitor disconnection if any were also noted. Statistical methods: Data was analyzed using

SUMMARY:
Compare haemodynamic changes and to evaluate the incidence of coughing, laryngospasm, loss of monitoring in patients undergoing lumbar disc surgery extubated in prone position and supine position.

DETAILED DESCRIPTION:
Tracheal irritation from the endotracheal tube, with subsequent coughing is common during emergence from general anaesthesia supine position and is often thought not to be a complication, but a physiological response to protect the airway from aspiration, although the side-effects of this vital reflex may be highly undesirable in clinical practice.

Coughing not only causes significant patient discomfort, but it may also cause hypertension, tachycardia, and increased intracranial, intraocular, and intra-abdominal pressure, which may lead to myocardial ischemia, arrhythmias, or surgical complications. Supine extubation also leads increased incidences of breath holding, laryngospasm, coughing, and monitor disconnection. These haemodynamic and airway responses are largely related movement of endotracheal tube during rolling of patients back to supine position during lighter depth of anaesthesia at conclusion of surgery. Coughing, breath holding, and laryngospasm also related to pooling of secretions to dependent patients airway in supine position.

Various techniques and drugs for the prevention of cardiovascular response and coughing during emergence have been studied, including extubation in a deep plane of anaesthesia, administration of intravenous drugs such as esmolol, lidocaine, short-acting opioids, or dexmedetomidine, and intracuff lidocaine. A reliable means of preventing undesired coughing has not been demonstrated to date.

Emergence in prone position has been found to be associated with less hemodynamic alterations, less coughing, laryngospasm, vomiting and monitor disconnections in patients undergoing lumbar surgery. There is a paucity of data regarding safety and efficacy of emergence from anaesthesia in prone position. The investigators present our initial experience of emergence from anaesthesia in prone position as compared to supine position in normotensive patients undergoing lumbar surgery in prone position.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-60 years
* prone surgery
* lumbar disc surgery

Exclusion Criteria:

* suspected difficult airway,
* risk factors for perioperative aspiration,
* chronic coughing,
* recent history of respiratory tract infection,
* chronic obstructive lung disease and
* obesity

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Heart rate changes from conclusion of surgery to extubation | From conlusion surgery to extubation of patient
  Heart rate and mean arterial pressure were recorded each minute till extubation Coughs, vomiting, laryngospasm and monitor disconnections were also recorded from conclusion of surgery (T0) till extubation.
Mean arterial pressure changes during emergence from anaesthesia | From conclusion of surgery to extubation
  Heart rate and mean arterial pressure were recorded each minute till extubation Coughs, vomiting, laryngospasm and monitor disconnections were also recorded from conclusion of surgery (T0) till extubation.

CONTACTS AND LOCATIONS:
Overall Officials: SHIVAKUMAR MC, MD, Principal Investigator — KVG Medical College and Hospital